CLINICAL TRIAL: NCT01829932
Title: The Effect of Prebiotics on the Microbiome in Irritable Bowel Syndrome Patients: The Diet and Microbiome Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Stephen Vanner, Professor of Medicine, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DMED-1443-11
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Diet
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Factor Diet (Active Comparator): Patients will be on a factor altered diet to see effects on their lactulose breath test and symptoms.
  Interventions: Dietary Supplement: Factor Altered Diet
- Low Factor Diet (Active Comparator): Patients will be on a factor altered diet to assess its effects on symptoms and lactulose breath test.
  Interventions: Dietary Supplement: Factor Altered Diet

INTERVENTIONS:
Dietary Supplement: Factor Altered Diet

SUMMARY:
Irritable bowel syndrome (IBS) is a chronic gastrointestinal illness of unknown cause whose symptoms include abdominal pain, bloating and altered bowel pattern. Diet has been shown to influence the bacteria gut interaction. Our aim is to determine if components of the diet affect IBS symptoms by changing the bacteria gut interaction. In particular, we will measure whether after being on a diet high or low on certain factors there is a change in the timing and amount of hydrogen and methane produced by bacteria digesting lactulose and on IBS symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Meet Rome III criteria for IBS
* Willing to undergo dietary intervention

Exclusion Criteria:

* History of Gastric, Small Bowel or Colonic Surgery
* History of Inflammatory Bowel Disease
* Celiac Disease
* Unable to come off following medications: antibiotics, laxatives, narcotics, sedatives
* On a pre specified diet
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area under the Curve of Hydrogen Gas on Lactulose Breath Test | 5 hours

SECONDARY OUTCOMES:
Change in Area Under the Curve on Lactulose Breath Test from Baseline | 5 hours
Change in IBS Symptom Severity Score from Baseline | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Vanner, MD, FRCPC, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] McIntosh K, Reed DE, Schneider T, Dang F, Keshteli AH, De Palma G, Madsen K, Bercik P, Vanner S. FODMAPs alter symptoms and the metabolome of patients with IBS: a randomised controlled trial. Gut. 2017 Jul;66(7):1241-1251. doi: 10.1136/gutjnl-2015-311339. Epub 2016 Mar 14. PMID 26976734